CLINICAL TRIAL: NCT01993706
Title: VRC 602: A Phase 1 Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIV MAB060-00-AB (VRC01),Administered Intravenously or Subcutaneously to Healthy Adults
Brief Title: Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC-HIVMAB060-00-AB (VRC01), Administered Intravenously or Subcutaneously to Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 140019; 14-I-0019
Record Dates: First submitted 2013-11-21; First posted 2013-11-25 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-02-27

CONDITIONS: HIV Infection; Monoclonal Antibody, Human; HIV Antibodies; VRC01 Monoclonal Antibody; Neutralizing Antibody
Keywords: Broadly HIV-1 Neutralizing Activity; Healthy Adults; Placebo; HIV Prevention; Monoclonal Antibodies; Antibodies
MeSH Terms: conditions — HIV Infections | interventions — VRC01 monoclonal antibody

INTERVENTIONS:
Drug: VRC-HIVMAB060-00-AB

SUMMARY:
Background:

- VRC01 is a manmade antibody directed against the human immunodeficiency virus (HIV). Antibodies fight infection. Researchers eventually want to know if VRC01 helps prevent or treat HIV infection. In this study they want to know if the study drug is safe if taken in a vein or under the skin. Taking VRC01 in this study will not protect against HIV infection.

Objectives:

- To see if VRC01 and placebo are safe and well tolerated.

Eligibility:

- Healthy adults 18 to 50 years old.

Design:

* Participants will be screened with medical history, physical exam, and lab tests.
* Participants will be randomly divided into 4 groups. VRC01 or the placebo will be given in weeks 1 and 4. Blood samples will be taken several times after each VRC01 or placebo dose.
* Three groups will receive VRC01 by needle into a vein with an IV pump. It will take about 1 hour and it is done in the hospital.
* One group will receive either VRC01 or the placebo by needle into the fatty tissue under the skin, usually the belly. It will take up to 20 minutes and it is done in the hospital.
* Participants will stay in the hospital overnight after receiving the medication and have about 14 clinic visits over 4 months. Most clinic visits last about 2 hours.
* Participants will keep a symptom diary after receiving the medicatino.
* Participants can volunteer to have mouth, rectal, and genital samples taken throughout the study.
* The study will last 8 months.

DETAILED DESCRIPTION:
Study Design: This is the first study in healthy adults of the VRC-HIVMAB060-00-AB (VRC01) monoclonal antibody (MAb). It is a dose-escalation study to examine safety, tolerability, dose, and pharmacokinetics of VRC01. The hypothesis is that VRC01 will be safe for administration to healthy adults by the intravenous (IV) and subcutaneous (SC) routes and will not elicit hypersensitivity reactions. A secondary hypothesis is that VRC01 will be detectable in human sera with a definable half-life. The SC route evaluation will be placebo-controlled and conducted double-blinded to evaluate safety and tolerability of VRC01 and placebo (VRC-PLAMAB068-00-AB).

Products Description: VRC-HIVMAB060-00-AB (VRC01) is a human MAb targeted to the HIV-1 CD4 binding site. It was developed by VRC/NIAID/NIH and manufactured under cGMP by the Vaccine Pilot Plant (VPP) operated by Leidos Biomedical Research, Inc. (formerly SAIC-Frederick, Inc.), Frederick, MD. Vials are provided at 100 plus or minus 10 mg/mL in a volume of 2.25 mL/vial.

VRC-PLAMAB068-00-AB (placebo) is a sterile, buffered aqueous solution of 25 mM Sodium Citrate, 50 mM Sodium Chloride, 150 mM L-Arginine Hydrochloride, 10% Dextran 40 (w/w), and 0.005% Polysorbate 80 (w/w) at pH 5.8. The placebo is filled at 2.25 plus or minus 0.1 mL/vial in 3 mL glass vials.

Subjects: Healthy adults, 18-50 years of age.

Study Plan: There are 3 open-label, dose escalation groups (Groups 1, 2, and 3) for IV administration and 1 blinded, placebo-controlled group (Group 4) for SC administration. Enrollment will start with subject randomization to Groups 1 and 4 in a 1:2 ratio. Within Group 4, subjects will be randomized to SC administration of VRC01 or placebo in a 1:1 ratio. No more than one subject per day in each group will receive the first IV infusion of the study product, and no more than one subject per week will receive the first SC infusion for the first 6 subjects in Group 4. If a first infusion is not administered or there are discontinuations from the study before there are sufficient data to conduct the dose escalation review for a group, then extra subjects may be enrolled into that group in order to have the requisite data on at least 3 subjects. Safety reviews of the IV Groups will be conducted 2 weeks after the third subject completes the Day 0 infusion. Safety review of Group 4 will be conducted 2 weeks after the sixth subject completes the Day 0 infusion.

After the IV dose escalation is complete, additional slots (up to 2 per schedule) may be filled in those schedules assessed as safe and well tolerated. The total accrual of 5 per schedule will provide additional safety and PK data to better inform product development. The additional enrollment slots will be filled by equal randomization of subjects to the 5 study schedules as they enroll. When completed with randomized enrollments, additional subjects may be enrolled and may receive a single VRC01 dose to evaluate the long-term pharmacokinetics.

Subjects will be admitted to an inpatient unit and remain for 24 hours following each product administration. Pharmacokinetic (PK) samples will be collected with each product administration at baseline and at specified intervals through 28 days after each product administration and at 56 days after the second product administration.

Due to the need to incur 3 days of disruption in normal daily activities that will begin with the first infusion, the enrollment day will most likely be different from Day 0. Safety lab samples will be collected at baseline, 2, 7, 14, and 28 days after each product administration. Subjects will keep a daily diary of solicited systemic symptoms for 3 days after each administration. Blood samples for human anti-VRC01 antibody evaluation will be drawn on Days 0, 14 and 56.

In all groups when the subject agrees, the oral and rectal fluid samples will be obtained at specified intervals after each product administration; women will also be offered cervical fluid sample collection.

Study Duration: The study is projected to take about 32 weeks to complete using the following assumptions:

* Individual subjects followed for 12 weeks after last VRC01 administration;
* All dosage groups completed;
* Enrollment of 3 subjects in the IV group per week during the IV dose escalation;
* Enrollments into Group 4 begin at the same time as Group 1.
* Additional subjects begin being randomized to all schedules assessed as safe and well tolerated beginning Week 16, and estimating 4 weeks to complete accrual and then 12 weeks to complete follow up of the last enrolled subject.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

1. Able and willing to complete the informed consent process.
2. 18 to 50 years of age.
3. Based on history and examination, must be in general good health without history of any of the conditions listed in the exclusion criteria.
4. Willing to have blood samples collected, stored indefinitely, and used for research purposes. [Note: Donation of mucosal samples is encouraged but not mandatory for eligibility.]
5. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
6. Screening laboratory values within 84 days prior to enrollment must meet the following criteria:

   * WBC 2,500-12,000/mm3
   * WBC differential either within institutional normal range or accompanied by the Principal Investigator or designee approval.
   * Platelets equal to 125,000 400,000/mm3
   * Hemoglobin within institutional normal range or accompanied by the Principal Investigator or designee approval.
   * Creatinine less than or equal to 1.1 x ULN
   * ALT less than or equal to 1.25 x ULN
   * Negative HIV serology

   FEMALE SPECIFIC CRITERIA:
7. If a woman is sexually active with a male partner and has no history of hysterectomy, tubal ligation or menopause, she must agree to use a prescription birth control method or a barrier birth control method from the time of study enrollment until the last study visit, or have a monogamous partner who has previously undergone a vasectomy.
8. Negative <=-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for women presumed to be of reproductive potential.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.
2. Weight >115 kg or <53 kg.
3. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence.
4. Hypertension that is not well controlled.
5. Woman who is breast-feeding, or planning to become pregnant during the 16 weeks of study participation.
6. Receipt of any investigational study agent within 28 days prior to enrollment or any past receipt of an investigational HIV vaccine.
7. Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer. Including, but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-11-19; Primary Completion 2015-02-27 (Actual); Study Completion 2015-02-27 (Actual)

PRIMARY OUTCOMES:
This is a Phase 1 study with primary outcomes of safety and pharmacokinetics | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wu X, Wang C, O'Dell S, Li Y, Keele BF, Yang Z, Imamichi H, Doria-Rose N, Hoxie JA, Connors M, Shaw GM, Wyatt RT, Mascola JR. Selection pressure on HIV-1 envelope by broadly neutralizing antibodies to the conserved CD4-binding site. J Virol. 2012 May;86(10):5844-56. doi: 10.1128/JVI.07139-11. Epub 2012 Mar 14. PMID 22419808
- [Background] Wu X, Yang ZY, Li Y, Hogerkorp CM, Schief WR, Seaman MS, Zhou T, Schmidt SD, Wu L, Xu L, Longo NS, McKee K, O'Dell S, Louder MK, Wycuff DL, Feng Y, Nason M, Doria-Rose N, Connors M, Kwong PD, Roederer M, Wyatt RT, Nabel GJ, Mascola JR. Rational design of envelope identifies broadly neutralizing human monoclonal antibodies to HIV-1. Science. 2010 Aug 13;329(5993):856-61. doi: 10.1126/science.1187659. Epub 2010 Jul 8. PMID 20616233
- [Background] Lynch RM, Tran L, Louder MK, Schmidt SD, Cohen M; CHAVI 001 Clinical Team Members; Dersimonian R, Euler Z, Gray ES, Abdool Karim S, Kirchherr J, Montefiori DC, Sibeko S, Soderberg K, Tomaras G, Yang ZY, Nabel GJ, Schuitemaker H, Morris L, Haynes BF, Mascola JR. The development of CD4 binding site antibodies during HIV-1 infection. J Virol. 2012 Jul;86(14):7588-95. doi: 10.1128/JVI.00734-12. Epub 2012 May 9. PMID 22573869
- [Derived] Ledgerwood JE, Coates EE, Yamshchikov G, Saunders JG, Holman L, Enama ME, DeZure A, Lynch RM, Gordon I, Plummer S, Hendel CS, Pegu A, Conan-Cibotti M, Sitar S, Bailer RT, Narpala S, McDermott A, Louder M, O'Dell S, Mohan S, Pandey JP, Schwartz RM, Hu Z, Koup RA, Capparelli E, Mascola JR, Graham BS; VRC 602 Study Team. Safety, pharmacokinetics and neutralization of the broadly neutralizing HIV-1 human monoclonal antibody VRC01 in healthy adults. Clin Exp Immunol. 2015 Dec;182(3):289-301. doi: 10.1111/cei.12692. Epub 2015 Sep 24. PMID 26332605